CLINICAL TRIAL: NCT00393562
Title: Comparison of Modafinil and Methylphenidate in Treatment of Excessive Daytime Sleepiness in Patients With Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit any subjects for this study
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Bucurescu, Gabriel - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PADRECC 01
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson's Disease
Keywords: excessive sleepiness; hypersomnolence; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Disorders of Excessive Somnolence | interventions — Modafinil; Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: modafinil
Drug: methylphenidate

SUMMARY:
This is an open-label cross-over randomized control study comparing the effect of modafinil and methylphenidate in patients with Parkinson's disease with excessive daytime sleepiness.

DETAILED DESCRIPTION:
Sleep disorders are common in Parkinson's disease (PD) and a significant cause of impairment of function in already disabled individuals. Almost all patients with PD report disturbed sleep, including excessive daytime sleepiness (EDS), disorders of initiating and maintaining sleep (DIMS) or parasomnias.1 The underlying pathology associated with PD and medication effects have both been implicated in the sleep disorders affecting these patients. EDS has become the focus of attention because of its effect on quality of life and impairment in driving and predisposition to traffic accidents. Its prevalence has been estimated between 15-50%. Treatment of EDS has become an important factor in the management of the PD patient, and the recent introduction of modafinil, a wakefulness promoting agent approved for narcolepsy, has led to increasing off-label use of this agent. Prior to modafinil, amphetamine and methylphenidate, two classical psychostimulants, were the agents of choice in treating EDS. However, these agents also have a direct effect on the dopaminergic system. They increase both sleep and REM latency, while reducing total sleep time and REM sleep. By comparison, the mechanism of action of modafinil is unknown, yet distinct from that of the psychostimulants. A direct comparison of the effect on EDS of modafinil with classical psychostimulants is lacking. The overall goals of this research proposal are to determine which agent is most effective in treating EDS in PD patients by using an open-label randomized control study comparing efficacy, onset of action and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Veteran at study site

Exclusion Criteria:

* Patients unable to give consent
* Diagnosis of EDS prior to diagnosis of PD
* Brain injury due to trauma, CVA, tumor or anoxia

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Compare efficacy of the two agents in treating excessive daytime sleepiness at 4 and 8 weeks

SECONDARY OUTCOMES:
Compare the safety profile of modafinil and methylphenidate

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Bucurescu, MD MS, Principal Investigator — Philadelphia, OPC
Locations (1):
- Philadelphia, OPC, Philadelphia, Pennsylvania, United States